CLINICAL TRIAL: NCT06362512
Title: An Innovative Cognitive-motor Exercise Training (COGMOTION) for People With Stroke: Effects on Balance, Mobility, Falls, Cognition and Related Brain Changes.
Brief Title: Cognitive-motor Exercise for Stroke Patients in Function, Cognition and Related Brain Changes.
Acronym: COGMOTION
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Marco_PANG_2024
Record Dates: First submitted 2024-04-08; First posted 2024-04-12 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-04

CONDITIONS: Stroke
Keywords: Dual-task training; Cognitive-motor interference
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: After stratification according to gender and walking speed, the participants will be randomly allocated to one of three groups: (1) dual-task training, (2) single-task training, and (3) control intervention, using a 1:1:1 allocation ratio.
Who Masked: Outcomes Assessor
Masking Description: This will be a single-blinded randomized controlled trial . The assessor will be blinded during assessments. The participants and investigators (trainers) are not possible to be blinded as it is an exercise intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- dual-task group (Experimental): patients receive three dual motor-cognitive exercise training per week for six weeks.
  Interventions: Behavioral: Dual-task training
- single-task group (Active Comparator): Patients receive three separate cognitive and mobility exercises per week for six weeks.
  Interventions: Behavioral: Single-task training
- control group (Active Comparator): Patients receive three upper limb muscle strengthening exercise with muscle stretching per week for six weeks.
  Interventions: Behavioral: Upper limb strengthening exercise

INTERVENTIONS:
Behavioral: Dual-task training — participants receive three 60-minute COGMOTION dual-task exercise sessions per week for six consecutive weeks.
  Arms: dual-task group
Behavioral: Single-task training — participants receive 30-minute single motor tasks with 30-minute single cognitive tasks three times per week for six consecutive weeks.The cognitive and mobility exercises will be the same as those in the dual-task group, but they will be performed separately.
  Arms: single-task group
Behavioral: Upper limb strengthening exercise — participants receive upper limb strengthening exercise for 30 minutes and flexibility exercises for 30 minutes three times per week for six consecutive weeks. The training is performed in sitting or standing position and no cognitive load will be added.
  Arms: control group

SUMMARY:
The purpose of this study is to evaluate a cognitive-motor exercise on dual-task interference during dual-task ankle movement and the corresponding alterations of brain activity.

DETAILED DESCRIPTION:
The prevalence rate of stroke increased by 106.0% (93.7-118.8) from 1990 to 2019 in China, and stroke burden is still severe. Community ambulation is an important factor that influences health-related quality of life after a stroke.In daily living, effective community ambulation requires the ability to maintain balance and walking function while engaging in other tasks that demand attentional resources simultaneously (i.e., dual-tasking). Increasing evidence has shown that stroke patients have more problems with dual-task balance and walking function than their age-matched able-bodied peers. stroke individuals were found to have more reduction in both the walking speed and cognitive recall than control group during walking with remembering a shopping list. Hence, since stroke victims must reintegrate into community, this kind of cognitive-motor interference needs to be thoroughly studied.

ELIGIBILITY:
Inclusion Criteria

Clinical diagnosis of stroke, Stroke onset of more than 6 months Aged 50 or more Capable of following verbal instructions Having a Montreal Cognitive Assessment score≥22, Able to walk for 1 minute without physical assistance Not receiving any formal rehabilitation training Having a Fugl-Meyer Ankle dorsiflexion-standing position score≥1

Exclusion Criteria

Contraindications to exercise (e.g., unstable angina) Contraindications to MRI (e.g., pacemaker) Color blindness Neurological disorders Gait-precluding pain Comorbidity

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-06-17 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Dual-task step frequency | before the initiation of training,after 6 weeks of training, 6 weeks after termination of the training
  step frequency under dual-task condition will be recorded
Dual-task cognitive performance accuracy | before the initiation of training,after 6 weeks of training, 6 weeks after termination of the training
  Number of correct responses will be measured during dual-task conditions

SECONDARY OUTCOMES:
Blood oxygenation level changes of the brain | before the initiation of training,after 6 weeks of training, 6 weeks after termination of the training
  Blood oxygenation level changes will be measured using Magnetic Resonance Imaging during dual-task conditions
Dual-task No.steps | before the initiation of training,after 6 weeks of training, 6 weeks after termination of the training
  No.steps under dual-task condition will be recorded
Dual-task correct reaction time | before the initiation of training,after 6 weeks of training, 6 weeks after termination of the training
  Correct reaction time under dual-task condition will be recorded
Dual-task amplitude of ankle movement | before the initiation of training,after 6 weeks of training, 6 weeks after termination of the training
  Amplitude of ankle movement under dual-task condition will be recorded

OTHER OUTCOMES:
Single-task walking speed | before the initiation of training,after 6 weeks of training, 6 weeks after termination of the training
  10-meter walking test will be used to assess single-task walking speed in meters per second
Dual-task walking performance | before the initiation of training,after 6 weeks of training, 6 weeks after termination of the training
  1 min Forward Walking with Serial 3 subtractions will be used to assess motor and cognitive performance during dual-task walking.
Mini Balance Evaluation Systems Test | before the initiation of training,after 6 weeks of training, 6 weeks after termination of the training
  Mini Balance Evaluation Systems Test will be used to assess postural control and balance, with total points from 0-28. Higher points indicate better performance.
Activities-specific Balance Confidence Scale | before the initiation of training,after 6 weeks of training, 6 weeks after termination of the training
  Activities-specific Balance Confidence Scale will be used to assess confidence of functional balance performance, with total points from 0-100. Higher points indicate better performance.
Trail Making Test | before the initiation of training,after 6 weeks of training, 6 weeks after termination of the training
  Trail Making Test will be used to assess executive function
Digit Span Test | before the initiation of training,after 6 weeks of training, 6 weeks after termination of the training
  Digit Span Test will be used to assess working memory
Montreal Cognitive Assessment | before the initiation of training,after 6 weeks of training, 6 weeks after termination of the training
  Montreal Cognitive Assessment will be used to assess global cognition, with total points from 0-30. Higher points indicate better performance.
Fall incidence | before the initiation of training, 6 months after training
  Monthly telephone interviews for recording fall incidence
Dual-task ankle movement degree | before the initiation of training,after 6 weeks of training, 6 weeks after termination of the training
  Ankle movement degree under dual-task condition will be recorded
Dual-task cognitive performance time | before the initiation of training,after 6 weeks of training, 6 weeks after termination of the training
  Time of correct responses under dual-task condition will be measured during dual-task conditions

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Yes
The study data can be provided via contacting the Principal Investigator
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From Dec 2026 onwards
Access Criteria: By contacting the Principal Investigator (Prof. Marco PANG): Marco.Pang@polyu.edu.hk